CLINICAL TRIAL: NCT07224204
Title: Life at 100.4: An Immersive Social Virtual Reality Education Tool for Adolescent and Young Adult Cancer Patients and Caregivers
Brief Title: Life at 100.4: An Immersive Social Virtual Reality (VR) Education Tool for Adolescent and Young Adult Cancer Patients and Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Glimpse Group Inc (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000040734; 1R41NR022239 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Adolescent Cancer; Young Adult Cancer
Keywords: Adolescent Cancer Patients and Caregivers; Young Adult Cancer Patients and Caregivers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: For Objective 1, an anticipated 20-30 participants for focus groups. For Objective 3, an anticipated 15 participant-caregiver-provider triads. Participants with new oncologic diagnosis and their caregivers at the Yale Pediatric Hematology/Oncology Clinic will be eligible for enrollment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Objective 1: Focus groups (No Intervention): Participants will participate in a 45 minute to 1-hour long focus group with similar stake holders to inform the intervention. These groups will take place via Zoom teleconferencing software, have 4-6 participants per group and will be run by appropriately trained study staff.
- Objective 3: (Experimental): Beta testing of VR-based educational intervention, Life at 100.4, to improve understanding of fever with neutropenia, how and when to check for it, and what to do when they have a fever.
  Interventions: Behavioral: Life at 100.4

INTERVENTIONS:
Behavioral: Life at 100.4 — An Immersive Social Virtual Reality Education Tool, participation up to 2 hours
  Arms: Objective 3:

SUMMARY:
The purpose of this study is to design and Beta test the Life at 100.4, an immersive social virtual reality education tool, with an anticipated 5 patient-caregiver-provider triads.Patients at Yale Pediatric Hematology and Oncology with a new oncologic diagnosis and their caregivers will be eligible for enrollment. Investigators will determine the feasibility and acceptability of implementing Life at 100.4 using validated measures.

DETAILED DESCRIPTION:
Febrile neutropenia, a condition marked by fever and low numbers of neutrophils, is the most commonly encountered complication of childhood cancer treatment. The mortality of untreated febrile neutropenia is as high as 30%. Delay of appropriate care and increased time to antibiotics are associated with increased mortality. Reasons for delay to care include a lack of understanding about the seriousness of febrile neutropenia or difficulty navigating the healthcare system. Effective, and evidence-based educational experiences can reduce morbidity and mortality rates related to febrile neutropenia. This proposal aims to combat knowledge gaps surrounding febrile neutropenia through the creation of an immersive social VR-based intervention, Life at 100.4. This program will provide critical education to patients and caregivers related to febrile neutropenia during cancer treatment. This work will result in the development of a critical new tool specific to febrile neutropenia while establishing VR more broadly as an effective patient and caregiver education tool, particularly for the near 40% of the population with low health literacy.

Objective 1 will include a qualitative study comprising interviews and focus groups with key stakeholders conducted by the Yale team to understand attitudes, perceptions, and knowledge around the navigation of febrile neutropenia.

Objective 2 will be the production of a VR-based prototype.

Objective 3, the focus of this registration, will assess feasibility and usability of this education tool.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with a malignancy or bone marrow failure condition
* Planned to receive chemotherapy and receive a central line

Exclusion Criteria:

* Medical contraindication to virtual reality including head wounds and history of seizure with flashing lights
* No plan to receive chemotherapy

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Multimodal Presence Scale for Virtual Environments | immediately post-intervention, up to 2 hours
  A 15-item validated tool to assess presence in VR. There are five items for each of the three dimensions, Physical Presence, Social Presence, and Self-Presence, scored on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree). Total score for each dimension 1-5 with higher scores indicating a stronger sense of presence in that dimension.
System Usability Scale (SUS) | immediately post-intervention, up to 2 hours
  A 10-item questionnaire with responses provided on a Likert scale. The SUS has been applied in evaluating the usability of different websites, software, and human computer interfaces. The final score is on a scale of 0-100. Higher scores indicate more usability.
Technology Acceptance Model (TAC) | immediately post-intervention, up to 2 hours
  Technology Acceptance Model questionnaire with questions related to Perceived Usefulness and Perceived Ease of Use. Total score range 1-5 with higher scores indicating higher acceptance and use.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Marks, MD, Principal Investigator — Yale University
Locations (1):
- Pediatric Hematology/Oncology Clinic in Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No